CLINICAL TRIAL: NCT01121159
Title: A Prospective Multicenter Study to Compare the Accuracy of Posttraumatic Orbital Reconstruction of the Medial Orbital Wall and/or the Orbital Floor With Preoperatively Preformed Versus Non-preformed Orbital Plates
Brief Title: Prospective Multicenter Trial to Compare Preformed vs Non Preformed Orbital Implants
Acronym: Orbita 3
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: Orbita3
Record Dates: First submitted 2010-05-07; First posted 2010-05-12 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Orbital Floor Fracture; Medial Orbital Wall Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preoperatively preformed orbital plates: Reconstruction with MatrixMIDFACE Preformed Orbital Plate (Synthes) or Custom-made orbital implant
  Interventions: Procedure: orbital fracture repair
- Non-preformed orbital plates: Reconstruction with Orbital Floor Mesh Plate or SynPOR Titanium Reinforced Fan Sheet (both Synthes)
  Interventions: Procedure: orbital fracture repair

INTERVENTIONS:
Procedure: orbital fracture repair — All patients will receive orbital fracture repair with one of the 4 specified implants

SUMMARY:
Accuracy of posttraumatic orbital reconstruction of the medial orbital wall and/or floor is better with preoperatively preformed orbital implants than with non-preformed orbital implants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years
2. Fracture (not older than 14 days) of the medial orbital wall and/or the orbital floor
3. Scheduled for reconstruction surgery with one of the following implants:

   * MatrixMIDFACE Preformed Orbital Plate
   * Custom-made orbital implant
   * Orbital Floor Mesh Plate
   * SynPOR Titanium Reinforced Fan Sheet
4. At least partial sight in both eyes before the accident
5. Willingness and ability to participate in the study follow-up according to the protocol
6. Ability to understand and read local language at elementary level
7. Signed informed consent

Exclusion Criteria:

1. Bilateral orbital fracture
2. Fractures of the orbital roof
3. Comminuted zygoma fracture
4. More than one piece fracture of the intraorbital bone lateral to the inferior orbital fissure
5. Previous dislocated orbital fractures on either side
6. Vision or diplopia not assessable
7. Injury of the globe
8. Neurological diseases with influence on eye motility or sight
9. Legal incompetence
10. Active malignancy
11. Life-threatening condition
12. Alcohol and drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with fractures of the orbital floor and/or medial orbital wall in one of the study centers
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
shape and volume assessing software | up to 3 days after surgery
  A post-op CT or CBCT scan will be analyzed with specially developed software that can compare shape and volume of the reconstruced orbit to the uninjured orbit.

SECONDARY OUTCOMES:
shape and volume assessing software | up to 3 days after surgery
  6 specific points and regions in the orbit will be compared between the reconstructed and the non-affected orbit
Clinical tests to assess vision | up to 3 days after surgery, 1 week after surgery, 4 weeks after surgery, 12 weeks after surgery
  Globe position, visual acuity, bulbus motility and diplopia will be assessed with clinical tests
Rate of complications | up to 3 days after surgery, 1 week after surgery, 4 weeks after surgery, 12 weeks after surgery
  Complications will be documented at every follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Niels Gellrich, Prof, Principal Investigator — Medizinische Hachschule Hannover
Locations (6):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Bundeswehrkrankenhaus Ulm, Ulm
- National University Hospital, Singapore, Singapore
- Hospital de 12 Octubre, Madrid, Spain

REFERENCES:
- [Result] Zimmerer RM, Ellis E 3rd, Aniceto GS, Schramm A, Wagner ME, Grant MP, Cornelius CP, Strong EB, Rana M, Chye LT, Calle AR, Wilde F, Perez D, Tavassol F, Bittermann G, Mahoney NR, Alamillos MR, Basic J, Dittmann J, Rasse M, Gellrich NC. A prospective multicenter study to compare the precision of posttraumatic internal orbital reconstruction with standard preformed and individualized orbital implants. J Craniomaxillofac Surg. 2016 Sep;44(9):1485-97. doi: 10.1016/j.jcms.2016.07.014. Epub 2016 Jul 21. PMID 27519662
- [Result] Zimmerer RM, Gellrich NC, von Bulow S, Strong EB, Ellis E 3rd, Wagner MEH, Sanchez Aniceto G, Schramm A, Grant MP, Thiam Chye L, Rivero Calle A, Wilde F, Perez D, Bittermann G, Mahoney NR, Redondo Alamillos M, Basic J, Metzger M, Rasse M, Dittman J, Rometsch E, Espinoza K, Hesse R, Cornelius CP. Is there more to the clinical outcome in posttraumatic reconstruction of the inferior and medial orbital walls than accuracy of implant placement and implant surface contouring? A prospective multicenter study to identify predictors of clinical outcome. J Craniomaxillofac Surg. 2018 Apr;46(4):578-587. doi: 10.1016/j.jcms.2018.01.007. Epub 2018 Feb 1. PMID 29530645
- See also: Link to published results — https://www.ncbi.nlm.nih.gov/pubmed/27519662
- See also: Link to published results — https://www.ncbi.nlm.nih.gov/pubmed/29530645